CLINICAL TRIAL: NCT06979102
Title: The Effect of Real Patient Interactive Stoma Care Management Teaching on Care Participation and Care Management Process of Ileostomy Patient and Caregiver: A Randomized Controlled Trial
Brief Title: The Effect of Real Patient Interactive Stoma Care Management Teaching
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Caz, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/10-28; 424S083 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye 1002-A Short Term Support Module)
Record Dates: First submitted 2025-04-27; First posted 2025-05-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-04

CONDITIONS: Ileostomy - Stoma; Caregiver; Care Management; Care Participation; Real Patient Interaction
Keywords: Caregiver; Ileostomy patient; Care management; Care participation; Real patient interaction; Teaching intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent researcher will perform randomization. She gave a signed document certifying her willingness to perform the randomization. Thus, the masking technique will be applied to the researchers until the implementation phase of the research starts. In the implementation phase of the research, masking won't be applied to ileostomy patients and their caregivers in the intervention and control groups. Also, one of the researchers and the stoma and wound care nurse won't be masked as they will be involved in the data collection phase. The other two researchers and the statistician who will perform the statistical analysis of the data will be masked until the analysis and interpretation phase of the research findings are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The real patient interactive stoma care management teaching will be carried out with ileostomy patients who have recently had their ileostomy opened and their caregivers in the intervention group.
  Interventions: Other: Real Patient Interactive Stoma Care Management Teaching
- Control Group (Active Comparator): The standard stoma care management teaching will be carried out with ileostomy patients who have recently had their ileostomy opened and their caregivers in the control group.
  Interventions: Other: Standard Stoma Care Management Teaching

INTERVENTIONS:
Other: Real Patient Interactive Stoma Care Management Teaching — The real patient interactive stoma care management teaching will be carried out with ileostomy patients who have recently undergone ileostomy surgery and their caregivers in the intervention group. The 2nd month after discharge, the newly ileostomy patients and their caregivers will be asked one open-ended question to elicit their thoughts and suggestions regarding the real patient interactive stoma care management teaching. The question is: "A real patient with a previous ileostomy participated in the stoma care management teaching. He demonstrated how to perform ileostomy care on himself and shared his experiences and suggestions regarding adapting to life with an ileostomy. What are your thoughts and suggestions regarding this teaching?"
  Arms: Intervention Group
Other: Standard Stoma Care Management Teaching — The standard stoma care management teaching will be carried out with ileostomy patients who have recently had their ileostomy opened and their caregivers in the control group.
  Arms: Control Group

SUMMARY:
Colorectal cancer is a type of cancer that is on the rise worldwide. Ileostomy with surgical treatment is one of the common treatment methods for this cancer. Regardless of whether the ileostomy is temporary or permanent, both patients with ileostomy and their caregivers are negatively affected physically and psychologically during this process. Patients with an ileostomy are especially at risk for ileostomy-related complications and metabolic complications. Stoma care management training on ileostomy care is critical in preventing these negativities. In this context, as a result of a real patient with ileostomy who has experience in opening an ileostomy and adapting to life with ileostomy, receiving structured training on stoma care teachings, the real patient with an ileostomy will take part in interactive stoma care management teachings in which the newly ileostomy patient and caregiver will take part together with a stoma and wound care nurses, and the processes of participation in care and care management of the newly ileostomy patient and caregiver will be improved, it is predicted that complications, physical and psychological problems that may develop related to ileostomy will be limited and contribute to public health in the long term. This research aims to determine the effect of real patient interactive stoma care management teaching on the processes of participation in care and care management of the newly ileostomy patient and caregiver. In this research, a randomized controlled full experimental research design with a post-test control group will be used. The population of the study will consist of newly ileostomy patients and their caregivers at Ankara Provincial Directorate of Health University of Health Sciences Gulhane Training and Research Hospital General Surgery Clinic. The sample of the study will be determined by using the criterion sampling method, one of the purposive sampling methods. Newly ileostomy patients and their caregivers who are eligible for the inclusion-exclusion criteria and who volunteer to participate in the study will be included. The research's data will be obtained using the Patient's Descriptive Characteristics Form, Caregiver's Descriptive Characteristics Form, Ostomy Self-Care Index, Caregiver Contribution to Self-Care in Ostomy Patient Index, Patient Health Engagement Scale, and Caregiver Health Engagement Scale. The implementation of the research will be carried out in two stages. In the first stage, real patients with an ileostomy will be identified, and training will be given to real patients on real patient interactive stoma care management with an ileostomy. In this context, to determine the expectations of individuals with stomas and their caregivers regarding stoma care management teaching, the plan was to determine the experiences of individuals with a prior permanent or temporary ileostomy/colostomy and current stomas and their caregivers regarding stoma care management education at the institution where the study was conducted. This plan was to structure the training to be delivered as part of the first stage of the study. To this end, ethics committee approval and institutional permission were obtained for the study titled "Determining the Stoma Care Education Experiences of Individuals with Stomas and Their Caregivers: A Qualitative Study." The opinions of individuals with stomas and their caregivers were collected, and the training was organized accordingly as part of the first stage of the study. In the second stage, real patient with ileostomy interactive stoma care management teaching will be applied to newly ileostomy patients and their caregivers in the intervention group, while standard stoma care management teaching will be applied to newly ileostomy patients and their caregivers in the control group. The objectives of this research are as follows: preparation of real patients with ileostomy; completion of real patients with ileostomy interactive stoma care management teaching with the intervention group; completion of standard stoma care management teaching with the control group; data analysis and statistical evaluations. It is predicted that with the real patient with ileostomy interactive stoma care management teaching, improvement will be achieved in the processes of participation in care and care management of the newly ileostomy patient and caregiver, complications, physical and psychological problems that may develop related to ileostomy will be limited, and in the long term, public health will be contributed.

ELIGIBILITY:
Inclusion Criteria:

For newly ileostomy patients;

* 18 years of age and over,
* Speak, read, write, and understand Turkish,
* Not having received teaching on stoma care and management before,
* No previous experience in stoma care and management. For caregivers;
* 18 years of age and over,
* Speak, read, write, and understand Turkish,
* Being an informal (unpaid) caregiver of a newly ileostomised patient,
* Not having received teaching on stoma care and management before,
* No previous experience in stoma care and management.

Exclusion Criteria:

For newly ileostomy patients; - Not participating in stoma care management teaching and follow-ups after ileostomy opening.

For caregivers;

- Not participating in stoma care management teaching and follow-ups after ileostomy opening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
To determine the processes of participation in care of the newly ileostomy patient with the Ostomy Self-Care Index | The second stoma care management teaching was completed before discharge, an average postoperative 6th day; The 2nd month after discharge.
  The scale has a 5-point Likert structure. The scale score is determined by adding the scores obtained from each item in the scale. As the scale score increases, the level of self-care management of the ostomy patient increases.
To determine the processes of participation in care of the caregiver with the Caregiver Contribution to Self-Care in Ostomy Patient Index | The second stoma care management teaching was completed before discharge, an average postoperative 6th day; The 2nd month after discharge.
  The scale has a 5-point Likert structure. The scale score is determined by adding the scores obtained from each item in the scale. As the scale score increases, the caregiver's support for the stoma-related self-care of the patient with an ostomy increases.
To determine the processes of care management of the caregiver with the Caregiving Health Engagement Scale | The second stoma care management teaching was completed before discharge, an average postoperative 6th day; The 2nd month after discharge.
  The scale has a total of 6 items and each item includes 4 statements and 7 options (A, B, C, D, E, F and G); options A and B are in the denial phase and have a score of 1, options C and D are in the hyperactivation phase and have a score of 2, options E and F are in the drowning phase and have a score of 3, option G is in the balance phase and has a score of 4; the scores of the caregiver for each item are ranked and the median value of the scores shows the participation phase in which the caregiver is located.
To determine the processes of care management of the newly ileostomy patient with the Patient Health Engagement Scale | The second stoma care management teaching was completed before discharge, an average postoperative 6th day; The 2nd month after discharge.
  The scale has a total of 5 items and each item contains 4 statements and 7 options (A, B, C, D, E, F and G); A and B options are in the blackout phase and have a score of 1, C and D options are in the arousal phase and have a score of 2, E and F options are in the adhesion phase and have a score of 3, G option is in the eudaimonic project and has a score of 4; the scores the patient receives for each item are listed and the median value of the scores shows the participation phase the patient is in.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Provincial Directorate of Health University of Health Sciences Gülhane Training and Research Hospital, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No